CLINICAL TRIAL: NCT01713699
Title: Determining the Sensitivity and Specificity of Circulating Tumor Cells and Cytology in Cerebrospinal Fluid of Patients Clinically Suspected for Leptomeningeal Metastases
Brief Title: Circulating Tumor Cells and Cytology in Cerebrospinal Fluid of Patients Clinically Suspected for Leptomeningeal Metastases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: N12CLM
Record Dates: First submitted 2012-10-22; First posted 2012-10-25 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Meningeal Carcinomatosis
Keywords: CTC, cytology, meningeal carcinomatosis, leptomeningeal metastases
MeSH Terms: conditions — Meningeal Carcinomatosis; Neoplastic Cells, Circulating | interventions — Spinal Puncture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- diagnostic (Other): Using extra CSF material received by clinically indicated lumbar punctures to determine the sensitivity and specificity of CTCs in CSF (5ml CSF). Standard material of 5 ml CSF for cytology and 2 ml CSF for cell count and chemistry is being regularly used and processed.
  Interventions: Procedure: lumbar puncture

INTERVENTIONS:
Procedure: lumbar puncture

SUMMARY:
The purpose of this study is to determine whether the quantitative detection of circulating tumor cells (CTCs) in patients with Epcam expressing tumors can be used compared to standard qualitative method - cytology both in the cerebrospinal fluid of patients, clinically suspected for leptomeningeal metastases.

DETAILED DESCRIPTION:
Leptomeningeal metastases (LM), is a diffuse dissemination of tumor cells into the cerebrospinal fluid (CSF) and leptomeninges.[1] Up to 8% of all patients with cancer develop LM. Gadolinium enhanced MRI of the symptomatic location of the nervous system is the radiological method of choice when LM is clinically suspected. In patients with a metastasized tumor, based on clinical signs of LM and contrast enhancement of either the leptomeninges, pia mater/cortex or cranial or spinal nerves on MRI, the diagnosis LM can be made. The sensitivity of MRI with gadolineum for LM is 75% and the specificity 77%. If MRI does not show equivocal abnormalities, CSF cytology needs to be performed. In 55% of patients with LM from solid tumors, malignant cells are found during the first CSF examination. The sensitivity raises to 80-90% after the second CSF sampling, as determined in the pre-MRI era. The volume of sampled CSF determines partly the sensitivity of CSF cytology. If possible, 10 ml CSF needs to be taken and the material must be processed as quickly as possible.

Recently, Patel et al (2011) described the detection of breast cancer cells in the CSF using the Cell Search System (Veridex). [6] Using this method, the CSF is enriched immuno-magnetically for the epithelial cell adhesion molecule (EpCAM). Next nuclear staining with 4 ',6-diamidino-2-phenylindole (DAPI) and immunofluorescent detection with cytokeratin and CD45 is performed in 5 patients with leptomeningeal metastases from breast cancer and approximately 104 circulating tumor cells (CTCs)in 7,5 ml CSF were found, using this method. There seemed to be an association between the number of CTCs and response to intrathecal administered chemotherapy in this small group of patients.

In the future, the determination of CTCs in the CSF could be a new quantitative method for the anti-tumor response assessment of systemic or intrathecal therapy (as opposed to CSF cytology, which is subjective and not a quantitative method). If the method shows greater sensitivity than CSF cytology and can reliably measure single tumor cells, the sensitivity of CSF examination in patients with a clinical suspicion of LM will increase. Possibly, this method can also be used to detect micrometastases in the CSF in patients without neurological symptoms, but with a high risk of CNS metastases.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are treated for advanced EpCam positive solid tumors (such as breast cancer, lung cancer, gastrointestinal cancer)
* Age >= 18 years;
* Able and willing to give written informed consent;
* WHO performance status (0, 1, 2, 3 or 4);
* Able and willing to undergo lumbar puncture and veni-puncture.

Exclusion Criteria:

* Lumbar puncture not clinically / diagnostically indicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2012-09; Primary Completion 2016-09-06 (Actual); Study Completion 2017-09-19 (Actual)

PRIMARY OUTCOMES:
Determine the sensitivity and specificity of detection of circulating tumor cells (CTCs) in patients with Epcam expressing tumors compared to cytology in the cerebrospinal fluid of patients, clinically suspected for leptomeningeal metastases | 3 months after end of study

SECONDARY OUTCOMES:
- To determine the relationship between the number of CTCs in CSF and the patient's neurological condition and WHO performance score | 3 months after end of study
- To determine the change in the CTC number between two sampling points and correlate this with the patient's neurological condition and therapy | 3 months after end of study
- To determine the relationships between demographics/tumor status and CTCs number in CSF. | 3 months after end of study
- To determine the relationship between the CTC cells in the CSF and the CTCs in the peripheral blood | 3 months after end of study
To confirm EPCAM positivity in archived primary tumor tissue and tumorcells in CSF. | 3 months after end of study
- To compare the predictive value of two CTC enumeration methods | 3 months after end of study

CONTACTS AND LOCATIONS:
Overall Officials: D. Brandsma, MD, PhD, Principal Investigator — NKI-AvL
Locations (2):
- Netherlands (2):
  - Dutch Cancer Institute - Antoni van Leeuwenhoek, Amsterdam
  - Slotervaart Hospital, Amsterdam

REFERENCES:
- [Derived] Milojkovic Kerklaan B, Pluim D, Bol M, Hofland I, Westerga J, van Tinteren H, Beijnen JH, Boogerd W, Schellens JH, Brandsma D. EpCAM-based flow cytometry in cerebrospinal fluid greatly improves diagnostic accuracy of leptomeningeal metastases from epithelial tumors. Neuro Oncol. 2016 Jun;18(6):855-62. doi: 10.1093/neuonc/nov273. Epub 2015 Nov 12. PMID 26566655
- See also: NKI-AVL — http://www.nki.nl/Research